CLINICAL TRIAL: NCT03062800
Title: Study of Thalidomide With First-line Chemotherapy and as Maintenance Treatment of Advanced Nonsquamous NSCLC With Epidermal Growth Factor Receptor Wild-Type or Unknown Mutation Status: A Multicenter, Randomized, Prospective Clinical Trial
Brief Title: Study of Thalidomide in Treatment of Advanced Nsclc (Dream-003)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dream-003
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Advanced Nsclc
Keywords: thalidomide; pemetrexed; nsclc; maintenance treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thalidomide; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P+Cisplatin/Carboplatin+T (Experimental): Induction therapy (Platinum based chemotherapy combined with antiangiogenic therapy 4-6 cycles):
  Pemetrexed + Platinum + Thalidomide [pemetrexed (500mg/m^2)+cisplatin(75mg/m^2)or carboplatin(AUC=5) on day 1 of 21-days cycle, ivgtt +thalidomide 100-200mg/d ,oral, qn ]
  Continue maintenance therapy (It is defined when a drug included in the induction treatment is used as maintenance .Patients who had not progressed during induction phase will be in this phase):
  Thalidomide 100mg/d ,oral, qn, until either disease progression or unacceptable toxicity.
  Interventions: Drug: Thalidomide; Drug: pemetrexed; Drug: cisplatin; Drug: carboplatin
- P+Cisplatin/Carboplatin (Experimental): Induction therapy ( Platinum based chemotherapy 4-6 cycles):
  Pemetrexed + Platinum [pemetrexed (500mg/m^2)+cisplatin(75mg/m^2)or carboplatin(AUC=5) on day 1 of 21-days cycle,ivgtt ]
  Maintenance therapy (It is defined when a drug included in the induction treatment is used as maintenance .Patients who had not progressed during induction phase will be in this phase):
  Pemetrexed (500mg/m^2) on day 1 of 21-days cycle, ivgtt.until either disease progression or unacceptable toxicity
  Interventions: Drug: pemetrexed; Drug: cisplatin; Drug: carboplatin

INTERVENTIONS:
Drug: Thalidomide — 100-200mg/d,oral ,qn
  Other Names: H32026128
  Arms: P+Cisplatin/Carboplatin+T
Drug: pemetrexed — (500mg/m^2) on day 1 of 21-days cycle,ivgtt
  Other Names: H20090232
Drug: cisplatin — (75mg/m^2) on day 1 of 21-days cycle, ivgtt
  Other Names: H20040813
Drug: carboplatin — (AUC=5) on day 1 of 21-days cycle, ivgtt
  Other Names: H20020180

SUMMARY:
The study for innovative strategies is warranted in the treatment of advanced non-squamous NSCLC with epidermal growth factor receptor wild-type or unknown mutation status because the outcomes remain unsatisfactory for most patients. Maintenance treatment after first-line chemotherapy is a very interesting strategy that has been largely investigated in the last years. This study is to evaluate the efficacy and toxicity of thalidomide in combination with chemotherapy and as maintenance treatment in patients with advanced non-squamous NSCLC.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer and is the leading cause of cancer mortality in the world. Every year, more than one million people die from lung cancer in worldwide. NSCLC accounts for about 85% of all lung cancers diagnosis and continues to remain a major therapeutic challenge.

Chemotherapeutic agents in the treatment of advanced NSCLC have reached a plateau of effectiveness when administered in the classic modality. In the first-line treatment of advanced non-squamous NSCLC with epidermal growth factor receptor wild-type, cisplatin plus pemetrexed is considered the best chemotherapeutic regimen. Recently, the PARAMOUNT trial has demonstrated that continuation maintenance with pemetrexed improves progression-free survival and overall survival after induction therapy with cisplatin plus pemetrexed in advanced non-squamous NSCLC with epidermal growth factor receptor wild-type.

Bevacizumab, a pure humanized anti-VEGF monoclonal antibody (mAb) has improved the outcomes of chemotherapy alone when combined with chemotherapy as first-line therapy for advanced non-squamous NSCLC. A randomized phase Ⅲ trial named Eastern Cooperative Oncology Group E4559 has demonstrated that concurrent bevacizumab with chemotherapy followed by maintenance bevacizumab in previously untreated patients with advanced non-squamous NSCLC is associated with an increase in overall survival.

In China, the cost of continuation maintenance with pemetrexed or bevacizumab is high in the current economic environment.

Thalidomide is much cheaper than pemetrexed and bevacizumab, and has been shown to have activity in numerous malignancies. Although the exact anti-tumor mechanism is unknown, thalidomide exhibits both immuno-modulating and anti-angiogenic effects. Based on potentially synergistic mechanisms of action, thalidomide has the potential to enhance the activity of conventional chemotherapy. Results from previously published small studies in which thalidomide was given concurrently with conventional chemotherapy and was continued as maintenance therapy suggest that thalidomide might be effective in the treatment of patients with small cell lung cancer and NSCLC. Study and evaluation the efficacy and toxicity of thalidomide in combination with chemotherapy and as maintenance treatment in patients with advanced non-squamous NSCLC with epidermal growth factor receptor wild-type is necessary.

ELIGIBILITY:
Inclusion Criteria:

1. stage Ⅳ non-squamous NSCLC with epidermal growth factor receptor wild-type or unknown mutation status confirmed by molecular biology and histology.
2. age 18-70 years.
3. Eastern Cooperative Oncology Group performance status of 0 or 1 and life expectancy greater than 3 months.
4. no previous treatment with chemotherapy or radiotherapy
5. adequate bone marrow, hepatic, and renal function
6. measurable or evaluable disease
7. informed consent
8. negative pregnancy test and adequate contraception for the duration of treatment

Exclusion Criteria:

1. malignancy during the 5 years previous to the diagnosis of NSCLC (unless nonmelanoma skin cancer or early cervical cancer)
2. surgery within 4 weeks
3. history of major hemoptysis
4. recent history of bleeding or thrombotic events
5. brain metastasis
6. uncontrolled hypertension
7. ongoing therapeutic anticoagulation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2 year
  Addition of thalidomide to chemotherapy and as single maintenance treatment is associated with similar PFS with Control Arm.

SECONDARY OUTCOMES:
objective response rate(ORR) | 2 years
  Response rates are similar in the two treatment groups
weight | 2 years
  Thalidomide can increase the weight of the patient
vascular endothelial growth factor (VEGF) VEGF | 1 year
  Thalidomide can decrease the level of VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Xiuwen Wang, MD.PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villa C, Cagle PT, Johnson M, Patel JD, Yeldandi AV, Raj R, DeCamp MM, Raparia K. Correlation of EGFR mutation status with predominant histologic subtype of adenocarcinoma according to the new lung adenocarcinoma classification of the International Association for the Study of Lung Cancer/American Thoracic Society/European Respiratory Society. Arch Pathol Lab Med. 2014 Oct;138(10):1353-7. doi: 10.5858/arpa.2013-0376-OA. Epub 2014 Feb 26. PMID 24571650
- [Background] Sandler A, Yi J, Dahlberg S, Kolb MM, Wang L, Hambleton J, Schiller J, Johnson DH. Treatment outcomes by tumor histology in Eastern Cooperative Group Study E4599 of bevacizumab with paclitaxel/carboplatin for advanced non-small cell lung cancer. J Thorac Oncol. 2010 Sep;5(9):1416-23. doi: 10.1097/JTO.0b013e3181da36f4. PMID 20686429
- [Background] Iwasaki A, Kuwahara M, Yoshinaga Y, Shirakusa T. Basic fibroblast growth factor (bFGF) and vascular endothelial growth factor (VEGF) levels, as prognostic indicators in NSCLC. Eur J Cardiothorac Surg. 2004 Mar;25(3):443-8. doi: 10.1016/j.ejcts.2003.11.031. PMID 15019676
- [Background] Gridelli C, Maione P, Rossi A. The PARAMOUNT trial: a phase III randomized study of maintenance pemetrexed versus placebo immediately following induction first-line treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small cell lung cancer. Rev Recent Clin Trials. 2013 Mar;8(1):23-8. doi: 10.2174/15748871112079990040. PMID 23259416
- [Background] Zhou S, Wang F, Hsieh TC, Wu JM, Wu E. Thalidomide-a notorious sedative to a wonder anticancer drug. Curr Med Chem. 2013;20(33):4102-8. doi: 10.2174/09298673113209990198. PMID 23931282
- [Background] Lee SM, James L, Buchler T, Snee M, Ellis P, Hackshaw A. Phase II trial of thalidomide with chemotherapy and as maintenance therapy for patients with poor prognosis small-cell lung cancer. Lung Cancer. 2008 Mar;59(3):364-8. doi: 10.1016/j.lungcan.2007.08.032. Epub 2007 Oct 24. PMID 17920723